CLINICAL TRIAL: NCT05672446
Title: Evaluation of the Effect of Standardized Child Patient Use on Preparing the Child for Process Skill; A Mix Method Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hulya ZENGIN, Assistant professor, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1234567
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Anxiety; Pediatric Nursing; Patient Simulation; Self Efficacy; High Fidelity Simulation Training
Keywords: experiental learning; anxiety; pediatric nursing; patient simulation; self efficiacy; high fidelity simulation training
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research was carried out using a convergent parallel design, which is a mixed method, which includes a randomized controlled study with a pretest-posttest control group, which is one of the quantitative research methods, and a phenomenological approach, one of the qualitative research designs.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 49 students in the experimental group experienced the ability to prepare a school-age child for the procedure with a simulation using standardized pediatric patients.
  Interventions: Other: simulation with standardized child patient
- Control (No Intervention): No attempt was made to the students in the control group.

INTERVENTIONS:
Other: simulation with standardized child patient — 49 students in the experimental group experienced the ability to prepare a school-age child for the procedure with a simulation using standardized pediatric patients. In the simulation, a school-aged child was used as the standard patient.
  Arms: Experimental

SUMMARY:
Background: Performing simulation applications using standardized patients provides realistic educational results that support critical thinking and learning, conducted using complex, effective communication scenarios.

Objective: This study was planned to evaluate the effect of the use of standardized pediatric patient practice in pediatric nursing education on the ability of nursing students to prepare the child for the procedure.

Method: The research was conducted using a convergent parallel design, which is a mixed method design. Ethics committee approval was obtained with the decision numbered 19/376 regarding the ethical suitability of the research. The sample of the study consists of 106 students. The students included in the study were given an introductory information form and the state trait anxiety scale and self-efficacy efficacy scale as pre-tests, and then the theoretical course "Preparing the child for the process according to age periods and communicating with the child patient" was explained. The students were divided into intervention and control groups by randomization. The students in the intervention group participated in the simulation application using standardized pediatric patients. Qualitative data were collected during the debriefing phase of the simulation and student satisfaction and self-confidence in learning scale was applied to the students in the intervention group. Before clinical practice, state trait anxiety scale, self-efficacy scale and perceived learning scale were applied as posttests. During the clinical practice, all students were evaluated in terms of their ability to prepare a real school-age child patient for the procedure.

DETAILED DESCRIPTION:
Background The use of high-fidelity simulation in healthcare education has emerged as a solution to address clinical experiences where patient, educational, or clinical setting limitations exist. Simulation, used to provide competence and competence in learning, is a technique or tool that attempts are made to create features of the real world. In the simulation performed using standardized patients; The patient or case study is portrayed by playing the role/scenario prepared with structured steps. Use of standardized/simulated patient in teaching; It contributes to the development of students' communication skills, history taking and physical examination skills. Training using standardized patients cannot be substituted for encountering real patients, but it is accepted as a practice that should be increased in a standard and integrative way. Simulation-based education is ideal for nursing education because it is an interactive method that can be used to help teach cognitive, psychomotor, or affective skills to individuals or groups of any skill or proficiency level. Simulation is a technique that can be used as a training method and/or research method. Simulation gives the opportunity to apply techniques that cannot be applied or tested, and provides realism and standardization. It is stated that it is beneficial to use in high-risk applications such as pediatric applications and where the probability of encountering students is low. For the child, the concept of illness and hospitalization include experiences that cause fear and discomfort. The hospital environment, healthcare professionals, materials and procedures create a sense of uncertainty for all children in the hospital. All procedures applied in the hospital affect the child physically, emotionally, behaviorally and cognitively. As a result, many behaviors such as fear, anxiety, anger, aggressive behaviors, impaired concentration, and rejection of further medical applications develop in the child. If children are not prepared before the procedure, they may become withdrawn, never speak or become aggressive due to the fear and anxiety they experience. This situation increases the psychological and physical pain and pain sensation of the child and complicates the work of the healthcare team. Preparation before the procedure, support during the procedure and follow-up after the procedure can help the child cope with invasive interventions. Nurses trying to provide sensitive care to the child should assume that every procedure applied to the child may be traumatic for the child.

The school-age child knows about infections and how they spread. The child in this period has a realistic perception about the disease, the cause of the diseases and their effects on the organs. The concept of the child's body parts and functions begins to develop. It is important to learn the child's knowledge about hospitalization and medical procedures and correct misunderstandings through play. Before the procedure, it is necessary to introduce himself to the child and allow the child to introduce himself. Parents should be encouraged to be with the child. All procedures and their reasons should be explained to the child without using medical terminology. The materials to be used during the procedure should be introduced to the child, and if possible, the process should be shown to the child on a toy or anatomical drawing. Giving the child the opportunity to ask questions about the procedure and answering their questions will reduce their anxiety. He should be allowed to choose as much as possible and his participation in the process should be encouraged. Before starting the procedure, the child's consent should be obtained and the child's privacy should be considered during the procedures. It is important to be rewarded or appreciated for the compliant behaviors displayed during the procedure.

Child health and diseases nursing is one of the fields where the use of simulation is most necessary, since pediatric patients are more likely to be harmed by medical errors. The use of children as standardized patients in medical education; It is not very common because the physical and mental development of children is incomplete and it is difficult to train children as standardized patients. However, despite the difficulties, it is very necessary to use children as standardized patients, to protect real patients from inappropriate experiences and to ensure patient safety. Clinical practice of child health and diseases nursing often causes feelings of fear and anxiety, and this reduces the performance of students. Alleviating these concerns can contribute to improving student performance and quality of care in the pediatric clinical setting.

Studies using children as standard patients are very limited. This study was planned to evaluate the effect of using children as standard patients on the child's ability to prepare for procedures in pediatric nursing education.

Method

Design This research was planned to evaluate the effect of the use of standardized pediatric patient practice in child health and diseases nursing education on the ability of nursing students to prepare the child for the procedure. The convergent parallel design, which is one of the mixed method designs in which quantitative and qualitative research methods are used together, was used in the research. The purpose of the convergent parallel design is to collect different but complementary data on the same topic in order to best understand the research problem.

Sample and arrangements The sample of the study consists of 106 students studying in the third year of a nursing faculty and taking the child health and diseases nursing course. The inclusion criteria of the study are as follows; Being a third year student at the faculty of nursing, taking the child health and diseases nursing course for the first time, being able to speak and understand Turkish, and giving consent to participate in the research. The exclusion criteria of the study are as follows; Being a foreign student, having taken the Child Health and Diseases Nursing course before, not accepting to participate in the research.

Ethical considerations Ethics committee approval was obtained with the decision numbered 19/376 regarding the ethical suitability of the study. The purpose of the study and the process were explained to the participants, confidentiality was assured, and they were given the freedom to withdraw from the study at any time. After the researchers explained the informed consent form, written consent was obtained from the participants. Numbers were used instead of real names to identify the participants, and the letter M was added to these numbers in the intervention group and the letter K in the control group.

Measuring tools

* Introductory features form The introductory characteristics form contains the sociodemographic data of the students and was prepared by the responsible researchers.
* Perceived learning scale The perceived learning scale was developed by Rovai et al. (2009). The Turkish validity and reliability of the scale was performed by Albayrak et al. in 2014. The scale consists of 9 items and has three factors. The level of participation of each item in the scale; Definitely false (1) and absolutely true (7). A score between 9 and 63 is obtained from the entire scale. The Cronbach's alpha value of the scale was found to be 0.83.
* Self-efficacy efficacy scale It was developed by Sherer et al. in 1982 to measure the individual's general self-efficacy-efficacy perception. The Turkish validity and reliability of the self-efficacy efficacy scale was performed by Gözüm et al. in 1999. The Cronbach's alpha value of the scale was calculated as 0.81. The scale is a 5-point Likert type scale consisting of 23 items. For each item, one of the options 1-"Does not describe me at all", 2-"Describes me a little", 3-"I am undecided", 4-"Describes me well", 5-"Describes me very well' is expected to be ticked. Thus, each individual can get a total score between the lowest 23 and the highest 115. A high total score from the scale indicates a high perception of general self-efficacy, and a low total score indicates a low perception of self-efficacy.
* Student satisfaction and self-confidence in learning scale The scale, which is widely used to measure students' attitudes and beliefs about simulation, was published by the National League for Nurses=NLN. The Turkish validity and reliability of the scale were performed by Karaçay et al. in 2017. It consists of two sub-dimensions, "satisfaction in learning" and "self-confidence", and a total of 13 items. The student satisfaction sub-dimension score is obtained from the sum of the scores of the 1st, 2nd, 3rd, 4th and 5th items. The self-confidence in learning sub-dimension score is obtained from the sum of the scores of the 6th, 7th, 8th, 9th, 10th, 11th, 12th and 13th items. The highest total score that can be obtained from the scale is 65, and the lowest is 13. The high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence. The Cronbach's alpha value of the scale was found to be 0.88.
* State trait anxiety scale The state trait anxiety scale was developed by Spielberger et al. It was translated into Turkish by Öner and Le Compte (1985) and its validity and reliability studies were carried out. The Cronbach Alpha internal consistency coefficient for the Trait Anxiety scale ranged from 0.83 to 0.87; It was found to be between 0.94 and 0.96 for the State Anxiety Inventory. There are 40 expressions in the scale that individuals can use to express their feelings. The first twenty of them measure the level of anxiety related to the situation and are scored by putting four options for each statement. These are: "Not at all" (1), "Somewhat" (2), "Many" (3), "Totally" (4).
* Skill checklist for preparing the school-age child for processing The skill checklist for preparing the school-age child for processing was created by the responsible researchers by reviewing the literature. For the content validity of the skill checklist, expert opinion was obtained from the faculty members of Health Sciences University, Gülhane Nursing Faculty, Department of Child Health and Diseases Nursing.

The skill checklist for preparing the school-age child for processing consists of 9 items. While evaluating the students, each applied item was marked and it was accepted that the student got a "1" point from that item. Accordingly, a student can get a minimum of "0" and a maximum of "9" points from the skill checklist. The Cronbach alpha value of the skill checklist for preparing the school-age child for processing was calculated as 0.83.

Developing Scenarios Two scenarios were used in the simulation application. The scenarios were prepared by the responsible researchers who were trained in simulation training. While preparing the content of the scenarios, it was necessary to choose a skill for preparing the pediatric patient for the procedure. Taking the opinions of the faculty members of the Department of Child Health and Diseases Nursing at the University of Health Sciences, Gülhane Nursing Faculty, it was decided to choose the skill of preparing the child for bloodletting, which is one of the skills that students have the most difficulty during clinical practice.

While developing the scenarios, simulation practice standards of the International Association for Clinical Simulation and Learning Nursing (INACSL) were taken into account.

Standardized Patient Education Two school-age children aged 7-12 years were used as standardized pediatric patients. Due to the absence of children enrolled in standardized patient programs in our country, standardized pediatric patients were selected voluntarily among the school-age children of the faculty members of the Faculty of Health Sciences Gülhane Nursing Faculty. Standardized pediatric patients and their parents were informed about the study before participating in the study and their written consent was obtained. Their parents were present during the education of the children and the execution of the simulation.

When a literature review was made, it was determined that in standardized patient practice, a person should undergo 4-8 hours of training after accepting to be a "standardized patient". A total of 8 hours of standardized patient education was conducted with standard pediatric patients, lasting 2 hours in 4 separate sessions.

Intervention The quantitative part of the study was conducted in a randomized controlled manner. Students were randomly divided into two groups. Students in the intervention group were included in a simulation using standardized pediatric patients. In the simulation application, 6 groups, 5 of which were 8 students and 1 of which were 9 students, participated in the application. Two standardized pediatric patients played the prepared scenarios by repeating them 3 times. A time of 10 minutes is planned for each simulation application. One student in the group communicated with the standardized pediatric patient, and the other students took part as observers. The simulation application was recorded with the video recording method and the students were allowed to watch themselves in the analysis session held after the simulation. In the last step of the study, all students went into clinical practice and during the clinical practice, each student was evaluated in terms of their ability to prepare the child for the procedure.

Data collection The two-hour course "Preparing the child for the procedure according to age periods and communication with the child patient" was given to the students who formed the universe of the research. State trait anxiety scale and self-efficacy efficacy scale were applied as pre-tests to all students who accepted to participate in the study. In the debriefing session, each of these questions was discussed with the students one by one. After the debriefing session was completed, a form containing the questions asked to them in the decoding session was given to the students and they were asked to write their answers. The written answers of the students constitute the data of the qualitative part of this research.

After the analysis session of the simulation, the students in the intervention group were applied the student satisfaction and self-confidence scale used in education with simulation.

After the completion of the simulation application, state trait anxiety scale, self-efficacy efficacy scale, and perceived learning scale were administered to all students in the intervention and control groups as post-tests.

Analysis of data In the qualitative part of this mixed method research, the written answers given by the students to the questions asked to them during the analysis phase were analyzed with the content analysis method, one of the qualitative data analysis methods. In this study, deductive content analysis method was used. Qualitative data were read repeatedly by the responsible researchers and the data in the text were coded under the categories of "doing, watching, feeling, thinking". The editing phase was completed by analyzing the data and placing them in the relevant categories. The reporting stage, which is the last step of the content analysis method, was completed with the presentation of the content analysis steps and findings.

IBM SPSS Statistics 23 package program was used for statistical calculations and analysis of the quantitative data of the research. Normality assumptions of numerical variables were examined with Kolmogorov Smirnov normality test. Relationships between two independent categorical variables were interpreted with Chi-square analysis. Differences between two independent groups (eg, control and intervention groups) were analyzed using the Independent Sample T Test for normally distributed variables and the Mann Whitney U test for non-normally distributed variables. The differences between two dependent numerical variables (pretest and posttest) were examined with the Dependent Sample T test. Statistical significance in the analyzes was interpreted at the p<0.05 level.

Theoretical framework The theoretical framework of this research is David A. Kolb's experiential learning theory. Kolb; He designed learning in the form of a circle in his experiential learning theory. There are four basic learning stages in this learning circle. These stages are; These are the "concrete experience" and "abstract conceptualization" stages, which show the conceptualization of experiences, and the "reflective observation" and "active experience" stages, which show the transformation of experiences. Written answers to the questions asked to the students during the analysis phase of the simulation were coded for the concepts of "feeling", "watching", "thinking" and "doing". These concepts form the categories of this qualitative research. Qualitative data were read repeatedly by the responsible researchers and the data in the text were coded under the categories of "doing, watching, feeling, thinking".

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd year student of Health Sciences University Gülhane Nursing Faculty
* To be taking the Child Health and Diseases Nursing course for the first time
* Agree to participate in the research
* Being a Turkish citizen and able to speak and understand Turkish

Exclusion Criteria

* Being a foreign student
* To have taken the Child Health and Diseases Nursing course before
* Refusing to participate in the research

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
checklist for preparing the school-age child for processing skill | 4 weeks
  The skill checklist for preparing the school-age child for processing was created by the responsible researchers by reviewing the literature (Ball et al., 2014; Conk, Başbakkal, Yılmaz, & Bolışık, 2013; Çavuşoğlu, 2013). For the content validity of the skill checklist, expert opinion was obtained from the faculty members of Health Sciences University, Gülhane Nursing Faculty, Department of Child Health and Diseases Nursing.
  The skill checklist for preparing the school-age child for processing consists of 9 items. While evaluating the students, each applied item was marked and it was accepted that the student got a "1" point from that item. Accordingly, a student can get a minimum of "0" and a maximum of "9" points from the skill checklist.

SECONDARY OUTCOMES:
The state trait anxiety scale | 3 weeks
  The state trait anxiety scale was developed by Spielberger et al. (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It was translated into Turkish by Öner and Le Compte (1985) and its validity and reliability studies were carried out. There are 40 expressions in the scale that individuals can use to express their feelings. The first twenty of them measure the level of anxiety related to the situation and are scored by putting four options for each statement. These are: "Not at all" (1), "Somewhat" (2), "Many" (3), "Totally" (4).
self efficacy scale | 3 weeks
  It was developed by Sherer et al. in 1982 to measure the individual's general self-efficacy-efficacy perception. (Sherer et al., 1982). The Turkish validity and reliability of the self-efficacy efficacy scale was performed by Gözüm et al. in 1999. (My Eye & Aksayan, 1999). The scale is a 5-point Likert type scale consisting of 23 items. For each item, one of the options 1-"Does not describe me at all", 2-"Describes me a little", 3-"I am undecided", 4-"Describes me well", 5-"Describes me very well' is expected to be ticked. Thus, each individual can get a total score between the lowest 23 and the highest 115. A high total score from the scale indicates a high perception of general self-efficacy, and a low total score indicates a low perception of self-efficacy.
perceived learning scale | 3 weeks
  The perceived learning scale was developed by Rovai et al. (2009) (Rovai, Wighting, Baker, & Grooms, 2009). The Turkish validity and reliability of the scale was performed by Albayrak et al. in 2014 (Albayrak, Güngören, & Horzum, 2014). The scale consists of 9 items and has three factors. The level of participation of each item in the scale; Definitely false (1) and absolutely true (7). A score between 9 and 63 is obtained from the entire scale.
Student satisfaction and self-confidence in learning scale | 1 weeks
  - Student satisfaction and self-confidence in learning scale The scale, which is widely used to measure students' attitudes and beliefs about simulation, was published by the National League for Nurses=NLN. (Franklin, Burns, & Lee, 2014). The Turkish validity and reliability of the scale were performed by Karaçay et al. in 2017. (Karaçay & Kaya, 2017). It consists of two sub-dimensions, "satisfaction in learning" and "self-confidence", and a total of 13 items. The highest total score that can be obtained from the scale is 65, and the lowest is 13. The high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya ZENGIN, Study Chair — Yuksek Ihtisas University
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No